CLINICAL TRIAL: NCT02888808
Title: Relationship Between Body Mass Index, Waist Circumference, Waist Hip Ratio and Erosive Gastroesophageal Reflux Disease in a Tertiary Centre in Nigeria: a Case Control Study
Brief Title: Relationship of Obesity With GERD Among Nigerians
Status: Completed | Type: Observational
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Olusegun Adekanle, Dr, Obafemi Awolowo University Teaching Hospital
Other Study IDs: ERC/2009/03/07
Record Dates: First submitted 2016-08-12; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Gastro-esophageal Reflux Disease With Ulceration.
Keywords: gastroesophageal reflux disease; women; Nigeria; obesity
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Erosive GERD: Gastroscopy examination.
  Interventions: Other: Gastroscopy
- Control population: Gastroscopy examination.
  Interventions: Other: Gastroscopy

INTERVENTIONS:
Other: Gastroscopy — Upper gastrointestinal endoscopy procedure

SUMMARY:
Obesity is a strong risk factor for GERD. This study assessed the role of obesity among patients having erosive GERD and controls.

DETAILED DESCRIPTION:
A case control study of patients with erosive GERD. Patients with erosive GERD who had upper gastro-intestinal endoscopy were graded using the Los Angeles classification. Patients and controls had measurements of body mass index (BMI), WC (waist circumference), Waist hip ratio (WHR), and hip circumference (HC). Bio-data was collected from both groups and data were analysed using descriptive and inferential statistics. A p value of equal to or less than 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyspepsia

Exclusion Criteria:

* Patients that refused consent.
* Patients with gastric cancer
* Patients with gastric outlet obstruction
* Pregnant women
* Active gastrointestinal bleeding
* Cigarette smokers
* Patients on Naso-gastric tube.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nigerians with dyspeptic symptoms
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Obesity associated with GERD | Immediate.
  Measurement of anthropometric indices

SECONDARY OUTCOMES:
Body mass index is associated with GERD | Immediate
  Measurement of body mass index (kilogram per meter squared)
Waist circumference is associated with GERD | Immediate
  Measurement of waist circumference (centimeter)
Waist hip ratio is associated with GERD | Immediate
  Measurement of waist hip ratio

IPD SHARING:
Plan to Share IPD: No